CLINICAL TRIAL: NCT03660033
Title: ECG Monitoring During NRP: a False Sense of Security?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Michael Andrew Assaad, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-2022
Record Dates: First submitted 2018-07-11; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Neonatal Resuscitation; Simulation
Keywords: Simulation; NRP; Resuscitation; ECG; Electrocardiogram
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: Participants will be invited to the mother-child simulation centre at CHU Sainte-Justine for a 60 minute simulation session during which they will complete two neonatal resuscitation scenarios (one of pulseless VT and the other of PEA). They will be randomized to either having access or not to ECG monitoring during the resuscitations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With ECG (Experimental): These teams will have access to ECG monitoring (intervention) during the scenario
  Interventions: Diagnostic Test: ECG in delivery room
- Without ECG (No Intervention): These teams will NOT have access to ECG monitoring during the scenario

INTERVENTIONS:
Diagnostic Test: ECG in delivery room — See arm/group discussions
  Arms: With ECG

SUMMARY:
ECG monitoring is relatively new mode of monitoring in the delivery room. While its use has been positively received by many practitioners of NRP, concerns have been raised about delaying chest compressions for a pulseless baby who may have electrical cardiac activity. It is unknown whether ECG leads do indeed provide a false sense of security in the delivery room. The investigators will be investigating this further using simulation.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether the presence of ECG monitoring has an impact on the resuscitative steps of NRP providers.

Participants will be invited to the mother-child simulation center at CHU Sainte-Justine for a 60 minute simulation session during which they will complete two neonatal resuscitation scenarios (one of pulseless VT and the other of PEA). They will be randomized to either having access or not to ECG monitoring during the resuscitations.

Investigators will plan to have participant teams perform the second scenario two weeks after the first scenario. This will be to hopefully mitigate repetition bias, as both scenarios will involve a pulseless newborn.

1. Resuscitation team and equipment Participants will be invited to be part of a three-person resuscitation team (physician or nurse practitioner, respiratory therapist and nurse) to complete the scenarios. A high-fidelity manikin will be utilized in all scenarios (Laerdal © Sim NewB). All necessary equipment as per NRP guidelines for neonatal resuscitation will be present at the bedside for the team to use.
2. Simulation scenarios In each group, the participants will be asked to proceed with the resuscitation of a newborn in the delivery room. Two different rhythms were chosen to see if changes seen with one abnormal appearing rhythm (ventricular tachycardia) can be replicated with a second normal appearing rhythm (PEA). Both of these rhythms cannot be considered normal as the newborn is pulseless.

   For the VT scenario, the newborn will be born in pulseless VT, with a pulse reading of 120 on the ECG monitor. There will have been an uneventful delivery. Participants will be expected to perform defibrillation, endotracheal intubation, chest compressions, umbilical venous catheter placement and intravenous epinephrine. Once the epinephrine is administered, the manikin will have a palpable pulse of 100, which will end the scenario.

   For the PEA scenario, the newborn will have a history of volume loss secondary to placenta previa. Because of the prolonged in utero asphyxia, the baby will be born in PEA arrest, with a heart rate display on the monitor of 80-90. In this scenario, resuscitative steps will include positive pressure ventilation, endotracheal intubation, chest compressions, umbilical venous catheter placement and intravenous epinephrine. Once the epinephrine is administered, the manikin will have a palpable pulse of 100, which will end the scenario.
3. Video recording of scenarios In order to be precise about time measurements, the investigators will record the resuscitations with the help of a video camera. The camera shot will only include the newborn manikin and the resuscitation team's hands. These recordings will not provide any identification data and will be for the sole purpose collecting data for this study. The video will be analyzed by the principal investigator and deleted in accordance with IRB guidelines.

The following data below will be collected. Please note that all time measurements will be from the start of the scenario.

* Time to pulse checks
* Time to application of ECG electrodes (for relevant scenarios)
* Number of subsequent pulse checks after application of ECG electrodes
* Method of pulse check (auscultation, palpation of the umbilical cord or brachial pulse)
* Time to start of chest compressions
* Time to administration of epinephrine

A questionnaire for each participant will collect the following data prior to the simulations: occupation, number of years of training in neonatology, number of years of experience in neonatology, last NRP course and approximate number of resuscitations in past year.

ELIGIBILITY:
Inclusion Criteria:

* Regular providers of neonatal resuscitation at our institution
* This includes residents, fellows, neonatal nurse practitioners, attending physicians, transport nurses and respiratory therapists
* Consents to the study (through a process of recruitment and informed consent)

Exclusion Criteria:

* Any individual who does not regularly participate in neonatal resuscitation in the delivery room
* Any individual who refuses consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Time to pulse check | 1 minute
  Time to pulse check once simulated manikin is programmed to be pulseless
Time to start of chest compressions | 2 minutes
  Time to start of chest compressions once simulated manikin is programmed to be pulseless
Time to administration of epinephrine | 3-4 minutes
  Time to administration of epinephrine once simulated manikin is programmed to be pulseless

SECONDARY OUTCOMES:
Number of subsequent pulse checks | 1-10 minutes
  After initial pulse check
Method of pulse check | 0-10 minutes
  Directly visualize (using video review) if participants use auscultation or palpation to check the pulse
Time of electrode placement | 0-10 minutes
  FOR ECG GROUP ONLY: time to application of ECG electrodes
Is the rhythm recognized? | 0-10 minutes
  FOR ECG GROUP ONLY: is the rhythm recognized Y/N?
Time to rhythm recognition | 0-10 minutes
  FOR ECG GROUP ONLY: measure at what time the team finally recognizes the baby's cardiac rhythm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali N, Sawyer T, Barry J, Grover T, Ades A. Resuscitation practices for infants in the NICU, PICU and CICU: results of a national survey. J Perinatol. 2017 Feb;37(2):172-176. doi: 10.1038/jp.2016.193. Epub 2016 Oct 27. PMID 27787506
- [Background] Fouzas S, Priftis KN, Anthracopoulos MB. Pulse oximetry in pediatric practice. Pediatrics. 2011 Oct;128(4):740-52. doi: 10.1542/peds.2011-0271. Epub 2011 Sep 19. PMID 21930554
- [Background] Hannibal GB. It started with Einthoven: the history of the ECG and cardiac monitoring. AACN Adv Crit Care. 2011 Jan-Mar;22(1):93-6. doi: 10.1097/10.1097/NCI.0b013e3181fffe4c. No abstract available. PMID 21297396
- [Background] Hay WW Jr, Rodden DJ, Collins SM, Melara DL, Hale KA, Fashaw LM. Reliability of conventional and new pulse oximetry in neonatal patients. J Perinatol. 2002 Jul-Aug;22(5):360-6. doi: 10.1038/sj.jp.7210740. PMID 12082469
- [Background] Jaeggi E, Ohman A. Fetal and Neonatal Arrhythmias. Clin Perinatol. 2016 Mar;43(1):99-112. doi: 10.1016/j.clp.2015.11.007. PMID 26876124
- [Background] Kamlin CO, Dawson JA, O'Donnell CP, Morley CJ, Donath SM, Sekhon J, Davis PG. Accuracy of pulse oximetry measurement of heart rate of newborn infants in the delivery room. J Pediatr. 2008 Jun;152(6):756-60. doi: 10.1016/j.jpeds.2008.01.002. Epub 2008 Mar 6. PMID 18492509
- [Background] Katheria A, Rich W, Finer N. Electrocardiogram provides a continuous heart rate faster than oximetry during neonatal resuscitation. Pediatrics. 2012 Nov;130(5):e1177-81. doi: 10.1542/peds.2012-0784. Epub 2012 Oct 22. PMID 23090347
- [Background] Kevat AC, Bullen DV, Davis PG, Kamlin CO. A systematic review of novel technology for monitoring infant and newborn heart rate. Acta Paediatr. 2017 May;106(5):710-720. doi: 10.1111/apa.13786. Epub 2017 Mar 6. PMID 28199732
- [Background] Wyllie J, Perlman JM, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2015 Oct;95:e169-201. doi: 10.1016/j.resuscitation.2015.07.045. Epub 2015 Oct 15. No abstract available. PMID 26477424
- [Background] Voogdt KG, Morrison AC, Wood FE, van Elburg RM, Wyllie JP. A randomised, simulated study assessing auscultation of heart rate at birth. Resuscitation. 2010 Aug;81(8):1000-3. doi: 10.1016/j.resuscitation.2010.03.021. Epub 2010 May 18. PMID 20483522
- [Background] Singh JK, Kamlin CO, Morley CJ, O'Donnell CP, Donath SM, Davis PG. Accuracy of pulse oximetry in assessing heart rate of infants in the neonatal intensive care unit. J Paediatr Child Health. 2008 May;44(5):273-5. doi: 10.1111/j.1440-1754.2007.01250.x. Epub 2007 Nov 12. PMID 17999668
- [Background] Maxwell LG, Harris AP, Sendak MJ, Donham RT. Monitoring the resuscitation of preterm infants in the delivery room using pulse oximetry. Clin Pediatr (Phila). 1987 Jan;26(1):18-20. doi: 10.1177/000992288702600102. PMID 3791833
- [Background] O'Donnell CP, Kamlin CO, Davis PG, Morley CJ. Feasibility of and delay in obtaining pulse oximetry during neonatal resuscitation. J Pediatr. 2005 Nov;147(5):698-9. doi: 10.1016/j.jpeds.2005.07.025. PMID 16291367
- [Background] Louis D, Sundaram V, Kumar P. Pulse oximeter sensor application during neonatal resuscitation: a randomized controlled trial. Pediatrics. 2014 Mar;133(3):476-82. doi: 10.1542/peds.2013-2175. Epub 2014 Feb 17. PMID 24534410
- [Background] Phillipos E, Solevag AL, Pichler G, Aziz K, van Os S, O'Reilly M, Cheung PY, Schmolzer GM. Heart Rate Assessment Immediately after Birth. Neonatology. 2016;109(2):130-8. doi: 10.1159/000441940. Epub 2015 Dec 19. PMID 26684743